Principal Investigator: John Corboy, MD

COMIRB No: 15-2388 Version Date: 10Jan2020

Study Title: Discontinuation of Disease Modifying Therapies (DMTs) in

Multiple Sclerosis (MS)

You are being asked to be in a research study. This form provides you with information about the study. A member of the research team will describe this study to you and answer all of your questions. Please read the information below and ask questions about anything you don't understand before deciding whether or not to take part.

# Why is this study being done?

Natural history research in MS suggests that risk of relapses and new Magnetic Resonance Imaging (MRI) changes diminishes significantly as people age, especially in MS patients 55 or older. Thus, the need to continue MS medicines that reduce relapses and new MRI lesions may also decrease as people age, especially in those who have not had relapses or MRI scan changes for prolonged times. This study plans to learn more about the safety of stopping MS medication in this population, as compared to continuing on the medication.

You are being asked to be in this research study because you are 55 or older, have MS without recent disease activity, and have been on a stable MS medication for the past 5 years.

## Other people in this study

Up to 60 people from your area will participate in the study.

Up to 265 people around the country will be in the study.

# What happens if I join this study?

This study will have 2 different groups of research subjects like you. One of these groups will stay on their current MS medication, and one group will discontinue their medication. To decide which group you will be in, we will use a method of chance. This method is like flipping a coin or rolling dice. This is called "randomization".

In order to participate in this study, you must be OK with being randomized to either group (regardless of which group you are assigned to, you and your doctor will make decisions about your medical treatment based on what is right for you, as explained later in this section).

If you join the study, you will be randomized to one of the 2 groups as described above. You will have some extra assessments done at you regular routine MS clinic appointment or at a separate research appointment today and every 6 months for the next 2 years, for a total of 5 visits. If you join the study after July 31, 2019, you may only complete 4 visits total. If you have a suspected relapse during these 2 years, we will also do these research procedures at your routine clinic visit or a separate research visit.

The following items will be done in addition to any assessments or procedures you are already having done as part of your clinical care and are the only items to be paid for by the study:

- Some questionnaires about your quality of life including questions about health, mood, thinking, and social life
- Some questionnaires about your MS symptoms
- A test of your attention, concentration, and thinking that involves numbers
- A test of your physical symptoms
- Along with the MRIs you get as part of your routine care, you will also have one 6
  months from today as part of the study. This 6 month MRI is the only MRI to be
  paid for by the study.
  - If you receive your routine MS care at an outside clinic, you should request to have standard MRIs once a year as part of your routine care while enrolled in this study and the results of these MRIs should be shared with the study team.

These things (not including the MRI) should take about an hour.

During months when you do not have the research procedures done, the study staff will call you to ask about changes in your health and potential relapses.

Regardless of which group you are assigned to, you and your doctor will make decisions about your medical treatment based on what is right for you. If new disease activity occurs or for other reasons, you and your doctor might decide to make changes to your therapy and you would no longer be able to be in your study "group". If this occurs, we would still like you to continue to complete the all the study procedures throughout the 2 years.

At the end of the study, you can decide whether or not to continue your current treatment strategy, and we will ask you what your decision is. This will occur prior to the overall results of the study being known. After the study results have been analyzed,

study personnel will contact you with the overall results. You and your doctor will make whatever decisions or changes about future medication use at that time.

We may also collect information from standard clinical MRIs you receive for up to 6 months after your last study visit.

## What are the possible discomforts or risks?

This trial is designed to evaluate the risks of 2 different treatment strategies (staying on MS drug vs. stopping MS drug). Each of these treatment strategies has possible risks.

- It is possible that stopping your MS medication may lead to an increase in disease activity.
- Continuing on your MS medication involves all of the risks of the drug itself, which should have been discussed with your as part of your clinical care.

In this study we will take Magnetic Resonance Images (MRI's) of your head. The MRI machine uses powerful magnetic waves to take pictures inside the body. The waves themselves are not harmful, but they can cause metal to heat up and electronics to stop working. You should NOT have an MRI if you have metal or electronic devices inside your body. Heart pacemakers and insulin pumps are examples of electronic devices. The MRI machine is a small round tube. It might make you uncomfortable if you do not like tight spaces. The most common side effect of having an MRI is flashing lights in the eyes. This is caused by the magnetic waves and is not harmful. Some people also experience warmth and reddening of the skin. This usually goes away after a few minutes.

Other possible risks include boredom or fatigue when completing the study assessments.

There is a risk that people outside of the research team will see your research information. We will do all that we can to protect your information, but it cannot be guaranteed.

The study may include risks that are unknown at this time.

## What are the possible benefits of the study?

This study is designed for the researcher to learn more about the risks of stopping MS medication.

This study is not designed to treat any illness or to improve your health. Also, there may be risks, as discussed in the section describing the discomforts or risks.

## Are there alternative treatments?

If you choose not to take part in the study, you can continue your current treatment or work with your doctor to discontinue your MS medications.

# Who is paying for this study?

This research is being funded by the Patient Centered Outcomes Research Institute and the National MS Society.

## Will I be paid for being in the study?

You will be paid \$40.00 for each of the 5 visits at which research procedures are completed. This will add up to a total of \$200 if you complete all of the study procedures at 5 visits. If you leave the study early, if you were enrolled after July 31, 2019, or if we have to take you out of the study, you will be paid only for the visits with research procedures that you have completed.

It is important to know that payments for participation in a study is taxable income.

## Will I have to pay for anything?

It will not cost you anything to be in the study. However, note that all procedures and assessments done as part of your routine clinical care, including MS drug, will be billed to you or your insurance per standard of care.

In addition, you may have increased costs (copays, hospitalizations, etc.) for treatment if your disease worsens during the study due to stopping MS medications.

## Is my participation voluntary?

Taking part in this study is voluntary. You have the right to choose not to take part in this study. If you choose to take part, you have the right to stop at any time. If you refuse or decide to withdraw later, you will not lose any benefits or rights to which you are entitled.

If there are any new findings during the study that may affect whether you want to continue to take part, you will be told about them.

# Can I be removed from this study?

The study doctor may decide to stop your participation without your permission if the study doctor thinks that being in the study may cause you harm, or for any other reason.

## What happens if I am injured or hurt during the study?

If you have an injury while you are in this study, you should call Dr. Corboy immediately. His phone number is 303-724-2187.

We will arrange to get you medical care if you have an injury that is caused by this research. However, you or your insurance company will have to pay for that care.

# Who do I call if I have questions?

The researcher carrying out this study is Dr. John Corboy. You may ask any questions you have now. If you have questions, concerns, or complaints later, you may call Dr. Corboy at 303-724-2187. You will be given a copy of this form to keep.

You may have questions about your rights as someone in this study. You can call Dr. Corboy with questions. You can also call the responsible Institutional Review Board (COMIRB). You can call them at 303-724-1055.

# Who will see my research information?

The University of Colorado Denver (UCD) and its affiliated hospital(s) have rules to protect information about you. Federal and state laws including the Health Insurance Portability and Accountability Act (HIPAA) also protect your privacy. This part of the consent form tells you what information about you may be collected in this study and who might see or use it.

The institutions involved in this study include

- University of Colorado Denver
- University of Colorado Hospital

We cannot do this study without your permission to see, use and give out your information. You do not have to give us this permission. If you do not, then you may not join this study.

We will see, use and disclose your information only as described in this form and in our Notice of Privacy Practices; however, people outside the UCD and its affiliate hospitals may not be covered by this obligation.

We will do everything we can to maintain the confidentiality of your personal information but confidentiality cannot be guaranteed.

The use and disclosure of your information has no time limit. You can cancel your permission to use and disclose your information at any time by writing to the study's Principal Investigator (PI), at the name and address listed below. If you do cancel your permission to use and disclose your information, your part in this study will end and no further information about you will be collected. Your cancellation would not affect information already collected in this study.

John Corboy, MD 12631 E. 17<sup>th</sup> Ave, mailstop B185 Aurora. CO 80045

Both the research records that identify you and the consent form signed by you may be looked at by others who have a legal right to see that information, such as:

- Federal offices such as the Food and Drug Administration (FDA) and the Office of Human Research Protections (OHRP) that protect research subjects like you.
- People at the Colorado Multiple Institutional Review Board (COMIRB)
- The study doctor and the rest of the study team
- Patient Reported Outcomes Institute and National MS Society, who are paying for this research study
- Officials at the institution where the research is conducted and officials at other institutions involved in this study who are in charge of making sure that we follow all of the rules for research

We might talk about this research study at meetings. We might also print the results of this research study in relevant journals. But we will always keep the names of the research subjects, like you, private.

You have the right to request access to your personal health information from the Investigator. To ensure proper evaluation of test results, your access to these study results may not be allowed until after the study is completed.

The investigator (or staff acting on behalf of the investigator) will use your information for the research outlined in this consent form. They will also make *all or some* of the following health information about you collected in this study available to:

- University of Alabama Birmingham (data coordinating center)
- Cleveland Clinic (central MRI reader)

# Information about you that will be seen, collected, used and disclosed in this study:

- Name and Demographic Information (age, sex, ethnicity, address, phone number, etc.
- Portions of your previous and current Medical Records that are relevant to this study, including but not limited to Diagnosis(es), History and Physical, laboratory or tissue studies, radiology studies, procedure results
- Research Visit and Research Test records

What happens to Data that are collected in this study?

Scientists at the University of Colorado Denver and the hospitals involved in this study work to find the causes and cures of disease. The data collected from you during this study are important to this study and to future research. If you join this study:

- The data given by you to the investigators for this research no longer belong to you.
- Both the investigators and any sponsor of this research may study your data collected from you.
- If data are in a form that identifies you, UCD or the hospitals involved in this study may use them for future research only with your consent or Institutional Review Board (IRB) approval.
- Any product or idea created by the researchers working on this study will not belong to you.
- There is no plan for you to receive any financial benefit from the creation, use or sale of such a product or idea.

# Agreement to be in this study and use my data

I have read this paper about the study or it was read to me. I understand the possible risks and benefits of this study. I understand and authorize the access, use and disclosure of my information as stated in this form. I know that being in this study is voluntary. I choose to be in this study: I will get a signed and dated copy of this consent form.

| Signature: | Date: |
|---|---|
| Print Name: | |
| Consent form explained by: | Date: |
| Print Name: | |
| Signature Line for witness; required for consent of non-reading subshort form | jects and consent using a<br>□ N/A |
| Witness Signature: | Date |
| Witness Print Name: | |
| Witness of Signature Witness of consent process | |